CLINICAL TRIAL: NCT02340806
Title: Effect of Epidural Infusion Bolus Delivery Rate on the Duration of Labor Analgesia
Brief Title: Association Between Bolus Rate and the Adequacy of Labor Analgesia Using Timed-intermittent Boluses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Elizabeth Lange, Assistant Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00100819
Record Dates: First submitted 2014-12-29; First posted 2015-01-19 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Labor Pain; Obstetric Pain
Keywords: epidural bolus; pain management; labor analgesia
MeSH Terms: conditions — Labor Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High rate bolus (CADD-Solis pump) (Experimental): Labor analgesia will be maintained using timed-intermittent boluses of local anesthetic with PCEA using the CADD-Solis pump. The bolus rate will be 300 mL/h in the high-rate bolus group.
  Interventions: Device: CADD-Solis pump (Smiths Medical)
- Low rate bolus (CADD-Solis pump) (Experimental): Labor analgesia will be maintained using timed-intermittent boluses of local anesthetic with PCEA using the CADD-Solis pump. The bolus rate will be 100 mL/h in the low-rate bolus group.
  Interventions: Device: CADD-Solis pump (Smiths Medical)

INTERVENTIONS:
Device: CADD-Solis pump (Smiths Medical) — The maintenance epidural solution for both groups will be bupivacaine 0.625 mg/mL with fentanyl 1.95 mcg/mL. The intermittent bolus volume will be 10 mL administered every 60 minutes. The first bolus will be given 30 minutes after intrathecal injection. In addition to the programmed boluses, patients will be able to administer patient-controlled epidural analgesia (PCEA) boluses of 5 mL every 10 minutes to a maximum of 15 mL (three PCEA boluses in a one hour period).

SUMMARY:
Administration of anesthetic solution into the epidural space is usually accomplished by a combination of continuous infusion, provider-administered boluses and patient-administered boluses (patient controlled epidural analgesia [PCEA]). The optimal method for maintaining labor analgesia is unknown. Several studies have demonstrated that timed-intermittent boluses, in combination with patient-controlled epidural analgesia (PCEA), provide superior maintenance of labor analgesia than maintenance with a continuous infusion with PCEA. Epidural infusion pumps capable of delivering timed boluses of local anesthetic with PCEA recently became commercially available. Several infusion rates are available for delivering the timed bolus, and the optimal bolus rate is unknown.

DETAILED DESCRIPTION:
Cervical dilation will be confirmed by a member of the obstetric team prior to epidural catheter placement as is routinely done at our institution. A baseline pain visual analog scale (VAS) score will be obtained using a 100-mm unmarked line with the end points labeled "no pain" and "worst pain imaginable.

Labor analgesia will be initiated using CSE analgesia with 25 mcg of intrathecal fentanyl. An epidural test dose will be performed as routine (1.5% lidocaine with epinephrine 1:200, 3 mL).

Labor analgesia will be maintained using timed-intermittent boluses of local anesthetic with PCEA using the CADD-Solis pump (Smiths Medical). An unblinded anesthesia research nurse will program the epidural pump and initiate the maintenance of labor analgesia.

Fifteen minutes following the intrathecal dose, a VAS score and a sensory level of analgesia will be obtained. The following information will be obtained hourly until complete cervical dilation (10 cm): VAS pain score, sensory level, a modified Bromage score (0 - no motor paralysis; 1 - inability to raise extended leg, but able to move knee and foot; 2 - inability to raise extended leg and to move knee, but able to move foot; 3 - inability to raise extended leg or to move knee and foot).

The time to the first request for supplemental analgesia will be recorded on the study data sheet. The time, type and volume of local anesthetic used, and VAS scores before and 15 minutes after the redose will be recorded.

All other clinical management will be as per routine, and study participation will not interfere with anesthetic or obstetric care. Anesthesiologists will manage breakthrough pain in the usual manner (assessment of stage of labor and extend/density of neuraxial blockade, followed by the appropriate maneuver to reestablish adequate analgesia).

Following delivery, the patient will be asked to give one final VAS score and her overall satisfaction with labor using a 100 mm unmarked line. Mode of delivery, as well as the duration of the 1st and 2nd stage of labor will be recorded by study personnel.

Patient Controlled Epidural Analgesia (PCEA) pump utilization data will be downloaded from epidural pumps after delivery. This will include the time to first PCEA request, the number of PCEA demands, the number of times that PCEA boluses were delivered, the total amount of local anesthetic consumed.

ELIGIBILITY:
Inclusion Criteria:

Term, nulliparous, English-speaking patients with singleton vertex pregnancies, who were 18 years or older, who presented to the Labor and Delivery Unit of Prentice Women's Hospital of Northwestern Memorial Hospital in spontaneous labor or for induction of labor were eligible to participate in the study

Exclusion Criteria:

History of chronic opioid analgesic use, prior opioid administration during labor, refusal of a vaginal examination prior to initiation of combined spinal-epidural (CSE) analgesia, or the presence of contraindications to neuraxial analgesia, such as coagulopathy or sepsis. Patients with cervical dilation > 5cm at the request for an epidural analgesia and women that were dilated > 5cm upon presentation to the labor and delivery unit were not approached for inclusion in the study; patients were excluded from the study after randomization if request for provider-administered supplemental bolus, or delivery, occurred within 90 minutes of intrathecal injection, or if there was a need for epidural catheter replacement during labor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lange, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong CA, Ratliff JT, Sullivan JT, Scavone BM, Toledo P, McCarthy RJ. A randomized comparison of programmed intermittent epidural bolus with continuous epidural infusion for labor analgesia. Anesth Analg. 2006 Mar;102(3):904-9. doi: 10.1213/01.ane.0000197778.57615.1a. PMID 16492849
- [Background] Lim Y, Sia AT, Ocampo C. Automated regular boluses for epidural analgesia: a comparison with continuous infusion. Int J Obstet Anesth. 2005 Oct;14(4):305-9. doi: 10.1016/j.ijoa.2005.05.004. PMID 16154735
- [Background] Chua SM, Sia AT. Automated intermittent epidural boluses improve analgesia induced by intrathecal fentanyl during labour. Can J Anaesth. 2004 Jun-Jul;51(6):581-5. doi: 10.1007/BF03018402. PMID 15197122
- [Background] Capogna G, Camorcia M, Stirparo S, Farcomeni A. Programmed intermittent epidural bolus versus continuous epidural infusion for labor analgesia: the effects on maternal motor function and labor outcome. A randomized double-blind study in nulliparous women. Anesth Analg. 2011 Oct;113(4):826-31. doi: 10.1213/ANE.0b013e31822827b8. Epub 2011 Jul 25. PMID 21788309
- [Background] Kaynar AM, Shankar KB. Epidural infusion: continuous or bolus? Anesth Analg. 1999 Aug;89(2):534. doi: 10.1097/00000539-199908000-00063. No abstract available. PMID 10439786
- [Background] Hogan Q. Distribution of solution in the epidural space: examination by cryomicrotome section. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):150-6. doi: 10.1053/rapm.2002.29748. PMID 11915061
- [Background] Wong CA, McCarthy RJ, Hewlett B. The effect of manipulation of the programmed intermittent bolus time interval and injection volume on total drug use for labor epidural analgesia: a randomized controlled trial. Anesth Analg. 2011 Apr;112(4):904-11. doi: 10.1213/ANE.0b013e31820e7c2f. PMID 21430035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 220 patients met inclusion criteria.
Period: Overall Study
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Started | 108 | 112
Completed | 102 | 108
Not Completed | 6 | 4
Not completed — Protocol Violation | 2 | 0
Not completed — epidural catheter replaced | 2 | 1
Not completed — history of chronic pain medication | 1 | 0
Not completed — re-dose < 90 min of CSE | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump) | Total
Number analyzed (Participants) | 102 | 108 | 210
Age, Continuous [Median (Full Range); unit: years] | 32 [29 to 33] | 31 [29 to 33] | 31 [29 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 108 | 210
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 86 | 79 | 165
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 13 | 19
Gestational Age (weeks) [Median (Full Range); unit: Weeks] | 40 [39 to 41] | 40 [39 to 41] | 40 [39 to 41]
Body Mass Index (kg/m2) [Median (Full Range); unit: (kg/m2)] | 29 [27 to 33] | 29 [27 to 31] | 29 [27 to 33]
Labor Type [Count of Participants; unit: Participants]
  Spontaneous Labor | 31 | 35 | 66
  Induction of Labor | 71 | 73 | 144
Cervical dilation at request for epidural (cm) [Median (Inter-Quartile Range); unit: centimeters] | 2 [2 to 3.5] | 2 [2 to 4] | 2 [2 to 4]
VAS (visual analog scale) [Median (Inter-Quartile Range); unit: units on a scale] — Visual Analog Scale is a scale used for pain where 0 equals no pain and 100 equals worse pain imaginable on a millimeter scale of 0-100.
  units on a scale | 75 [63 to 87] | 73 [62 to 84] | 74 [62 to 86]
Mode of delivery [Count of Participants; unit: Participants] — Mode of delivery of the baby (vaginal delivery, assisted vaginal delivery or Cesarean delivery)
  Participants
    Vaginal Delivery | 69 | 71 | 140
    Assisted Vaginal Delivery | 9 | 13 | 22
    Cesarean Delivery | 24 | 24 | 48
Indication for Cesarean delivery [Count of Participants; unit: Participants] — Population: 24 participants in each group underwent cesarean section. The below analyzes the reason for cesarean section in each group.
  Participants
    number analyzed (Participants) | 24 | 24 | 48
    Arrest of dilation | 7 | 14 | 21
    Arrest of descent | 8 | 5 | 13
    Fetal Intolerance | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Breakthrough Pain.
Description: Number of participants who experienced breakthrough pain requiring a provider administered bolus by the anesthesia providers.
Time Frame: epidural placement to delivery, up to 36 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
Participants | 37 | 43
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .67, Chi-squared, Corrected

2. Secondary Outcome: Total Bupivacaine Consumption Per Hour of Labor Analgesia
Description: Total bupivacaine amount (milligrams/hour mg/h) via pump and provider administered supplemental boluses
Time Frame: epidural placement to delivery, up to 36 hours.
Measure: Median (Inter-Quartile Range); unit: milligrams per hour
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
milligrams per hour | 9.9 [8.1 to 11.4] | 10.8 [8.6 to 11.4]
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .08, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Number of Requested PCEA Boluses
Description: Number of PCEA (Patient Controlled Epidural Anesthesia) bolus doses delivered
Time Frame: epidural placement to delivery, up to 36 hours.
Measure: Median (Inter-Quartile Range); unit: Doses
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
Doses | 14 [6 to 27] | 17 [10 to 31]
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .21, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Total Number of Delivered PCEA Boluses
Description: Total number of PCEA (Patient Controlled Epidural Anesthesia) bolus's delivered.
Time Frame: epidural placement to delivery, up to 36 hours.
Measure: Median (Inter-Quartile Range); unit: Doses
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
Doses | 9 [5 to 18] | 10 [7 to 17]
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .14, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Ratio of Total Number of PCEA Boluses Requested and Delivered
Description: The ratio of the total number of PCEA (Patient Controlled Epidural Anesthesia) bolus's requested and PCEA doses delivered.
Time Frame: epidural placement to delivery, up to 36 hours.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
Ratio | 1.4 [1.2 to 2.1] | 1.5 [1.2 to 2.1]
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .66, Kruskal-Wallis

6. Secondary Outcome: Satisfaction Scores
Description: Patients overall satisfaction with pain management. The scale 0= poor satisfaction and 100= good satisfaction with pain management.
Time Frame: up to 24 hours after delivery
Measure: Median (Inter-Quartile Range); unit: score on a scale (0 poor 100 good)
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
score on a scale (0 poor 100 good) | 98 [86 to 100] | 98 [88 to 100]

7. Other Pre Specified Outcome: Time to Provider Administered Supplemental Boluses
Description: Time to provider administered supplemental boluses measured in minutes
Time Frame: epidural to first request of redose up to 10 hours
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
Minutes | 357 [215 to 525] | 302 [148 to 559]
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .92, Wilcoxon (Mann-Whitney)

8. Other Pre Specified Outcome: Mean Pain Score
Description: Weighted mean pain score (measured by the area under the VAS (Visual Analog Scale)-time curve calculated using the trapezoidal integration divided by the duration of labor analgesia).Visual Analog Scale is a 100 millimeter scale where 0 is no pain and 100 is worst pain imaginable.
Time Frame: epidural placement to delivery, up to 36 hours.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
units on a scale | 9 [3.9 to 17.2] | 6.9 [3.7 to 15]
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .58, Kruskal-Wallis

9. Other Pre Specified Outcome: Stage of Labor at Re-dose Request
Description: The stage of labor ( first or second) at the time of re-dose request.
Time Frame: Through 2 stages of labor up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
Participants
  First stage of labor | 34 | 40
  Second stage of labor | 3 | 3
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .67, Chi-squared

10. Other Pre Specified Outcome: Number of Participants With Epidural Re-doses
Description: Total number of patients requiring epidural re-doses given by the provider.
Time Frame: epidural placement to delivery, up to 36 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
Participants
  No- redoses | 59 | 71
  1 re-dose | 31 | 27
  2 re-doses | 6 | 5
  3 re-doses | 6 | 5
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .99, Chi-squared

11. Other Pre Specified Outcome: Patient Satisfaction of Labor Anesthesia
Description: Patient satisfaction of labor anesthesia using a score of 0 low satisfaction to 100 high satisfaction on a 100 millimeter scale.
Time Frame: Up to 24 hours after delivery of baby
Measure: Median (Inter-Quartile Range); unit: score on a scale (0 poor 100 good)
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
Number analyzed (Participants) | 102 | 108
score on a scale (0 poor 100 good) | 98 [86 to 100] | 98 [88 to 100]
Statistical Analysis 1: Comparison: High Rate Bolus (CADD-Solis Pump) vs Low Rate Bolus (CADD-Solis Pump); Test type: Superiority; p = .37, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 24 hours after delivery of the baby
Arm/Group | High Rate Bolus (CADD-Solis Pump) | Low Rate Bolus (CADD-Solis Pump)
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/108
Other Adverse Events (participants affected / at risk) | 0/102 | 0/108

LIMITATIONS AND CAVEATS:
Limiting our study subjects to nulliparous patients in early labor could have led to a cohort that was more prone to sysfunctional labor and these results could be different in multiparous women with shorter labors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT02340806/Prot_SAP_000.pdf